CLINICAL TRIAL: NCT01625585
Title: LONG-TERM OUTCOMES AFTER SINGLE-BALLOON ENTEROSCOPY IN PATIENTS WITH OBSCURE GASTROINTESTINAL BLEEDING
Brief Title: Single Balloon Enterosocpy Obscure Gastrointestinal Bleeding Bleed
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: SBEWashU 2012
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Obscure Gastrointestinal Bleeding
Keywords: Push-and-Pull Enteroscopy; Single-Balloon-Enteroscopy

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Consecutive patients undergoing SBE for OGIB

SUMMARY:
The goal of the present study is to investigate the clinical outcomes of patients with gastrointestinal bleeding originating from the small intestine following diagnostic investigation with single balloon enteroscopy. We hypothesize that single balloon enteroscopy can arrive at a diagnosis and provide therapeutics in a majority of patients with gastrointestinal bleeding originating in the small intestine.

DETAILED DESCRIPTION:
The small intestine has been, until recent years, a black box to gastroenterologists because it is difficult to see and reach. Radiological imaging provides little details of small intestinal mucosa. Capsule endoscopy, introduced in 2001, enables gastroenterologists to visualize the entire small intestine from within for the first time, but it is only a diagnostic tool. Single-balloon enteroscopy (SBE) is a new enteroscopy methods that use an overtube with one balloon or a spiral to help pleat bowel onto the endoscope and allow examination of the distal small bowel. This methods allow for biopsy, hemostasis, and other therapeutic interventions to be performed in the small bowel. Early reports have been promising; with 50-70% diagnostic yield for small bowel pathology reported in the literature. However, despite these promising results the impact SBE findings on patient outcomes is not clear.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Obscure Gastrointestinal Bleeding undergoing SBE at Barnes Jewish Hospital

Exclusion Criteria:

* Less than 3 months of follow up after SBE
* The endoscope could not be advanced into the duodenum will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent SBE at Washington University Medical Center/ Barnes Jewish Hospital prior to 1/1/2011 were eligible for inclusion. There was no control group as this was a retrospective cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Recurrence of obscure gastrointestinal bleeding following single balloon enteroscopy | 4 years
  The primary outcome is recurrence of gastrointestinal bleeding, defined as recurrent overt or occult gastrointestinal bleeding, hospitalization for gastrointestinal bleeding or acute blood loss anemia.

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital/ Washington University, St Louis, Missouri, United States